CLINICAL TRIAL: NCT01633385
Title: Lung Function and Bronchial Inflammation in Patients With Bronchiolithis Obliterans
Brief Title: Bronchial Inflammation in Patients With Bronchiolithis Obliterans
Acronym: FRABO-02
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: BO2012-02
Record Dates: First submitted 2012-06-26; First posted 2012-07-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Bronchiolitis Obliterans
Keywords: bronchial inflammation; Bronchiolitis obliterans; Sputum; Blood; Inflammation; adaptive immune system; innate immune system
MeSH Terms: conditions — Bronchiolitis Obliterans; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, sputum cells, sputum supernatans
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject-Group: Patients suffering from doctors diagnosed bronchiolitis obliterans
- Control Group: age- and sex matched to subject-group

SUMMARY:
The investigators plan to study the variability of lung function parameters and bronchial inflammatory markers in 20 patients with bronchiolitis obliterans at the age of 6 to 25 years compared with an age- and sex-matched control group. The investigators will perform a pulmonary function test (body plethysmography with TLCO), and measure the fraction of exhaled nitric oxide (eNO). Further a blood sample is drawn to determine the systemic inflammation. Finally induced sputum is collected and a cell count is performed, and cells and supernatants are analyzed for inflammatory markers. This investigation will be repeated after 4-6 weeks. The aim of this study is to define baseline values and the variability of possible outcome parameters for future interventional studies.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the variability of lung function values and bronchial inflammation of 20 Patients with Bronchiolitis obliterans aged between 6 up to 25 years. The patients' data will be compared with the results of a reference group with similar age conditions to determine possible outcome-parameters for following interventional studies.

The sputum samples will be processed and quantitatively analyzed to get a profile of the cytological composition.

(Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction (PCR) (qRT-PCR) and by cytometric bead assay (CBA).)

Methods and Work Programme:

This study consists of two study visits (V1 and V2)

V1:

* Measurement of nitric oxide in expired air (eNO)
* Lung function testing with spirometry and body plethysmography
* Bronchodilation
* Lung function testing with spirometry and body plethysmography
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, (genetic markers of the non-specific pulmonary defense system)
* Induced sputum for inflammatory mediators and microbiological investigations

V2:

* Measurement of nitric oxide in expired air (eNO)
* Lung function testing with spirometry and body plethysmography
* Bronchodilation
* Lung function testing with spirometry and body plethysmography
* Induced sputum for inflammatory mediators and microbiological investigations

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 6 and 25 years of age
* Known Bronchiolitis obliterans

  * no Bronchiolitis obliterans(depending on the study group)
* Ability to perform lung function tests and inhalation

Exclusion Criteria:

* Acute illness with systemic or bronchial inflammation
* every chronic condition or infection (eg HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study
* Participation in another study

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients suffering from Bronchiolitis obliterans and controls
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of FEF75 over time | V1: Day 1 - V2: Day 28-42
  Look for changes/ variability of this lung function parameter

SECONDARY OUTCOMES:
change of sputum cell count over time | V1: Day 1 - V2: Day 28-42
  induced sputum will be analyzed for different cellular components such as alveolar macrophages, neutrophils, lymphocytes and others. Epithelial cells will be excluded
change of low CrP over time | V1: Day 1 - V2: Day 28-42
  serum parameter for systemic inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Kurland G, Michelson P. Bronchiolitis obliterans in children. Pediatr Pulmonol. 2005 Mar;39(3):193-208. Review — http://www.ncbi.nlm.nih.gov/pubmed/15635614
- See also: Smith KJ, Fan LL. Insights into post-infectious bronchiolitis obliterans in children. Thorax. 2006 Jun;61(6):462-3. — http://www.ncbi.nlm.nih.gov/pubmed/16738042
- See also: Pichler M, Herrmann G, Schmidt H, Ahrens P, Zielen S. Persistent adenoviral infection and chronic obstructive bronchitis in children: is there a link? Pediatr Pulmonol. 2001 Nov;32(5):367-71. — http://www.ncbi.nlm.nih.gov/pubmed/11596161
- See also: Pichler MN, Reichenbach J, Schmidt H, Herrmann G, Zielen S. Severe adenovirus bronchiolitis in children. Acta Paediatr. 2000 Nov;89(11):1387-9. — http://www.ncbi.nlm.nih.gov/pubmed/11106056